CLINICAL TRIAL: NCT05209022
Title: Acute Effects of Beetroot Juice Ingestion on Components of Vertical Jump Performance
Brief Title: Beetroot Juice Ingestion and Vertical Jump Performance
Acronym: BEET_JUMP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad Francisco de Vitoria (Other)
Collaborators: Ankara University (Other); University of Seville (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Universidad_Francisco_Vitoria
Record Dates: First submitted 2022-01-14; First posted 2022-01-26 (Actual); Last update posted 2022-01-26 (Actual); Status verified 2022-01

CONDITIONS: Dietary Supplements

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Quadruple (Participant, Care Provider, Investigator, Outcomes Assessor)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Beetroot supplementation (Experimental): One serving 140 mL of beetroot juice (12.8 mmol of NO3-; Beet-It-Pro Elite Shot, James White Drinks Ltd., Ipswich, UK) after an overnight fast and 3 h before initiating the testing session.
  Interventions: Dietary Supplement: Beetroot juice
- Placebo supplementation (Placebo Comparator): One serving of beetroot juice depleted in NO3- (0.08 mmol of NO3-) as placebo (Beet It; James White Drinks Ltd, Ipswich, UK) after an overnight fast and 3 h before initiating the testing session.
  Interventions: Dietary Supplement: Beetroot juice

INTERVENTIONS:
Dietary Supplement: Beetroot juice — 140 mL of beetroot juice or beetroot juice placebo

SUMMARY:
Beetroot juice is a dietary supplement with good evidence for improving sports performance in different sport contexts, however, the evidence about the effects of beetroot juice in jump capacity is unclear. Thus, the aim of this study was to conduct a comprehensive examination of beetroot juice effects on vertical jump performance

DETAILED DESCRIPTION:
Beetroot juice is a dietary supplement with good evidence for improving sports performance in different sport contexts, however, the evidence about the effects of beetroot juice in jump capacity is unclear. Therefore a deeper knowledge about the effects of beetroot juice on several components of vertical jump performance remain largely unexplored between we can mention phase duration peak power, average power, peak velocity, initial force, and peak force. Thus, the aim of this study was to conduct a comprehensive examination of beetroot juice effects on several countermovement jump components.

ELIGIBILITY:
Inclusion Criteria:

Experience in resistance training (at least 18 months of three weekly sessions).

A one-repetition maximum weight (1 RM) higher than bodyweight in the bench press and of 1.5 of body weight in squat exercise No sports supplement was taken in the previous three months No smoking. No cardiovascular, pulmonary or neurological disease. To not be considered an elite athlete.

Exclusion Criteria:

Age <18 year or > 35 years.

Ages: 18 Years to 35 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Enrollment: 19 (Actual)
Dates: Start 2019-05-20 (Actual); Primary Completion 2019-06-20 (Actual); Study Completion 2019-06-20 (Actual)

PRIMARY OUTCOMES:
Jump height | 72-hours
  Maximal jump height using a force platform
Peak Power | 72-hours
  Maximal peak power obtained using a force platform
Average power | 72-hours
  Average power obtained using a force platform

SECONDARY OUTCOMES:
Peak velocity | 72-hours
  Peak velocity obtained using a force platform
Phase durations | 72-hours
  Concentric /Isometric/Eccentric phases obtained using a force platform

CONTACTS AND LOCATIONS:
Locations (1):
- Universidad Francisco de Vitoria, Madrid, Spain

IPD SHARING:
Plan to Share IPD: No